CLINICAL TRIAL: NCT01010919
Title: A Phase I Study of Chicory for Treatment of Osteoarthritis of the Hip or Knee
Brief Title: A Study of Chicory for Treatment of Osteoarthritis of the Hip or Knee
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Phytomedics Inc. (Industry)
Collaborators: University of Texas, Southwestern Medical Center at Dallas (Other)
Other Study IDs: PMI-005-01
Record Dates: First submitted 2009-11-06; First posted 2009-11-10 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

INTERVENTIONS:
Dietary Supplement: Chicory root extract

SUMMARY:
Extracts of chicory root have anti-inflammatory properties in vitro and in animal models of arthritis. The primary objective of this investigator-initiated, Phase 1, placebo-controlled, double blind, dose-escalating trial is to determine the safety and tolerability of a proprietary bioactive extract of chicory root in patients with osteoarthritis (OA). Secondary objectives are to assess effects on the signs and symptoms of this disorder. Individuals greater than 50 years of age with OA of the hip or knee will be eligible for trial entry.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 50 years of age or older and may be of either gender.
2. Patients must have have an imaging-confirmed (radiograph or MRI) diagnosis of OA of the hip or knee.
3. Patients must not have taken a nonsteroidal anti-inflammatory medication for at least 7 days prior to the baseline visit (a single daily aspirin 325 mg or less is allowed throughout the study).
4. Patients must be able and willing to give informed consent.

Exclusion Criteria:

1. Any unstable comorbid medical condition that in the opinion of the investigator could interfere with the ability of the patient to complete the study.
2. Patients who are unable to ambulate and require a wheelchair due to the severity of the arthritis are excluded. Ambulatory aids such as canes and walkers are acceptable.
3. Patients requiring continuing therapy with nonsteroidal anti-inflammatory drugs are excluded.
4. Patients requiring any dose of glucocorticoids within the past 30 days are excluded.

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult

REFERENCES:
- [Derived] Olsen NJ, Branch VK, Jonnala G, Seskar M, Cooper M. Phase 1, placebo-controlled, dose escalation trial of chicory root extract in patients with osteoarthritis of the hip or knee. BMC Musculoskelet Disord. 2010 Jul 9;11:156. doi: 10.1186/1471-2474-11-156. PMID 20618964